CLINICAL TRIAL: NCT02434250
Title: Effectiveness of Selective Laser Trabeculoplasty (SLT) After Failed Phacoemulsification Cataract Extraction Combined With Eximer Laser Trabeculectomy (Phaco-ELT) in Open Angle Glaucoma and Ocular Hypertension
Brief Title: Selective Laser Trabeculoplasty After Failed Phacoemulsification With Eximer Laser Trabeculectomy
Acronym: SLT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SLT after Phaco-ELT
Record Dates: First submitted 2015-01-29; First posted 2015-05-05 (Estimated); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: Open Angle Glaucoma; Ocular Hypertension; Cataract
Keywords: Open angle glaucoma; Ocular hypertension; Cataract; Selective Laser Trabeculoplasty; Eximer Laser Trabeculectomy; Phacoemulsification Cataract Extraction
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension; Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SLT arm (Experimental): Patient receiving 'Selective Laser Trabeculoplasty' (SLT) due to failed Phacoemulsification Cataract Extraction with Intraocular Lens Implantation combined with Eximer Laser Trabeculectomy (phaco-ELT) in Open Angle Glaucoma and Ocular Hypertension to control intraocular pressure and/or glaucoma progression.
  Interventions: Procedure: Selective Laser Trabeculoplasty

INTERVENTIONS:
Procedure: Selective Laser Trabeculoplasty — Selective Laser Trabeculoplasty is a laser treatment procedure to enhance trabecular aequous humor outflow and thus decrease intraocular pressure.

SUMMARY:
The aim of this study is to evaluate the efficacy of selective laser trabeculoplasty after a prior failed phacoemulsification and Eximer Laser Trabeculectomy.

DETAILED DESCRIPTION:
This study evaluates the efficacy of selective laser trabeculoplasty after a failed combined procedure of phacoemulsification cataract extraction with intraocular lens implantation plus Eximer Laser Trabeculectomy in open angle glaucoma or ocular hypertension. The success of SLT will be determined by the intraocular pressure and number of hypotensive drugs.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of open angle glaucoma or ocular hypertension
* and diagnosis of cataract

Exclusion Criteria:

* diagnosis of angle closure glaucoma
* any optic neuropathy other than glaucoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2015-05; Primary Completion 2016-10 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Efficacy intraocular pressure | t0 and t=12 month
  Efficacy as measured by decrease in intraocular pressure from baseline
Efficacy medication | t0 and t=12 month
  as measured by decrease in number of used hypotensive medications

SECONDARY OUTCOMES:
Efficacy visual acuity | t0 and t=12 month
  Efficacy as increase in best corrected visual acuity

CONTACTS AND LOCATIONS:
Overall Officials: Marc Toeteberg-Harms, MD, FEBO, Principal Investigator — UniversityHospital Zurich, Dept. of Ophthalmology
Locations (1):
- Department of Ophthalmology, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No